CLINICAL TRIAL: NCT06187597
Title: Efficacy and Safety of Toripalimab After Concurrent Chemoradiotherapy in Elderly Patients With Esophageal Squamous Cell Carcinoma: a Multicenter, Randomized, Phase II Trial (EC-CRT-007)
Brief Title: Consolidation of Toripalimab After Chemoradiotherapy in Elderly Esophageal Cancer (EC-CRT-007)
Acronym: EC-CRT-007
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); Zhujiang Hospital (Other); Fifth Affiliated Hospital, Sun Yat-Sen University (Other); Xiangya Hospital of Central South University (Other); Wuhan University (Other)
Responsible Party: Principal Investigator, Mian XI, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2023-503
Record Dates: First submitted 2023-12-16; First posted 2024-01-02 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Locally Advanced Esophageal Squamous Cell Carcinoma
Keywords: Esophageal squamous cell carcinoma; Chemoradiotherapy; Immunotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — S 1 (combination); Tegafur; gimeracil; potassium oxonate; toripalimab; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The study group (Experimental): Patients will receive radiotherapy with prescribed dose of 54 Gy in 27 fractions, concurrently with S-1 chemotherapy. Then patients in the study group will receive toripalimab as consolidation therapy for up to 12 months (16 cycles) after the completion of chemoradiotherapy.
  Interventions: Drug: S-1; Drug: Toripalimab; Radiation: Intensity-modulated radiotherapy
- The control group (Active Comparator): Patients will receive radiotherapy with prescribed dose of 54 Gy in 27 fractions, concurrently with S-1 chemotherapy. Then patients will be receive routine follow-up.
  Interventions: Drug: S-1; Radiation: Intensity-modulated radiotherapy

INTERVENTIONS:
Drug: S-1 — Patients received S-1 administration, 70mg/m2 per day, orally on days 1 to 14 and 29 to 42 during radiotherapy.
  Other Names: Tegafur,Gimeracil and Oteracil Potassium Capsules
Drug: Toripalimab — Patients received toripalimab 240 mg every 3 weeks for up to 16 cycles.
  Other Names: Toripalimab Injection
  Arms: The study group
Radiation: Intensity-modulated radiotherapy — All patients received external-beam radiation using intensity-modulated radiotherapy. The prescribed dose is 54 Gy in 27 fractions over 5-6 weeks.
  Other Names: IMRT

SUMMARY:
Although definitive chemoradiotherapy (CRT) is the standard treatment option for unresectable locally advanced esophageal cancer, elderly patients tolerate intravenous concurrent CRT less well with age and comorbidities. Previous trials have demonstrated that CRT with oral S-1 was tolerable and provided significant survival benefits over radiotherapy alone in elderly patients with esophageal squamous cell carcinoma (ESCC). However, as high as 54% of patients with elderly ESCC experienced locoregional or distant recurrence after CRT. Therefore, a more effective regimen for older patients is needed. Immune checkpoint inhibitors targeting PD-1/PD-L1 have shown substantial clinical benefits in advanced esophageal cancer. Recently, the combination of immunotherapy with CRT has emerged as a promising strategy to improve clinical outcomes in locally advanced esophageal cancer. The aim of this study was to evaluate the efficacy and safety of toripalimab (an anti-PD-1 antibody) after concurrent CRT in elderly patients with locally advanced ESCC.

DETAILED DESCRIPTION:
A total of 140 patients with elderly, unresectable, locally advanced ESCC will be stratified according to age (70-80 vs. ≥80) and TNM stage (I/II vs. III/IV) and randomly assigned (1:1) to receive toripalimab as consolidation therapy for up to 12 months (arm A) or not (arm B) after definitive radiotherapy with concurrent S-1.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed squamous cell carcinoma of the esophagus;
2. Locally advanced, and absence of hematogenous metastasis disease according to UICC TNM version 8;
3. Not suitable for surgery (either for medical reasons or patient's choice);
4. Age at diagnosis 70 to 85 years;
5. No prior cancer therapy;
6. Estimated life expectancy >6 months;
7. Eastern Cooperative Oncology Group performance status ≤ 2
8. No history of concomitant or previous malignancy;
9. The function of important organs meets the following requirements: a. white blood cell count (WBC) ≥4.0×109/L, absolute neutrophil count (ANC) ≥1.5×109/L; b. platelets ≥100×109/L; c. hemoglobin ≥9g/dL; d. serum albumin ≥2.8g/dL; e. total bilirubin ≤1.5×ULN, ALT, AST and/or AKP ≤2.5×ULN; f. serum creatinine ≤1.5×ULN or creatinine clearance rate >60 mL/min;
10. Ability to understand the study and sign informed consent.

Exclusion Criteria:

1. Patients who have been treated previously with anti-tumor therapy (including chemotherapy, radiotherapy, surgery, immunotherapy, etc.);
2. Patients with hematogenous metastasis disease or esophageal fistula at diagnosis;
3. Known or suspected allergy or hypersensitivity to monoclonal antibodies, any ingredients of cadonilimab, and the chemotherapeutic drugs paclitaxel or cisplatin;
4. Patients who have a preexisting or coexisting bleeding disorder;
5. Inability to provide informed consent due to psychological, familial, social and other factors;
6. Presence of CTC grade ≥2 peripheral neuropathy;
7. A history of malignancies other than esophageal cancer before enrollment, excluding non-melanoma skin cancer, in situ cervical cancer, or cured early prostate cancer
8. A history of diabetes for more than 10 years and poorly controlled blood glucose levels;
9. Patients who cannot tolerate chemoradiotherapy due to severe cardiac, lung, liver or kidney dysfunction, or hematopoietic disease or cachexia.
10. Active autoimmune diseases, a history of autoimmune diseases (including but not limited to these diseases or syndromes, such as colitis, hepatitis, hyperthyroidism), a history of immunodeficiency (including a positive HIV test result), or other acquired or congenital immunodeficiency diseases, a history of organ transplantation or allogeneic bone marrow transplantation;
11. A history of interstitial lung disease or non-infectious pneumonia;
12. A history of active pulmonary tuberculosis infection within 1 year or a history of active pulmonary tuberculosis infection more than 1 year ago but without formal anti-tuberculosis treatment;
13. Presence of active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL), hepatitis C (positive for hepatitis C antibody, and HCV-RNA levels higher than the lower limit of the assay).

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From date of enrollment until the date of death from any cause or the date of first documented disease progression whichever came first, assessed up to 36 months.
  Three-year follow-up from the date of enrollment to the date of disease progression or last follow-up

SECONDARY OUTCOMES:
Overall survival | From date of enrollment until the date of death from any cause or the date of last follow-up, whichever came first, assessed up to 36 months.
  Three-year follow-up from the enrollment to the date of death from any cause or date of lost follow-up
Clinical complete response | 13-16 weeks after the completion of radiotherapy
  Tumor response was evaluated 13-16 weeks after the completion of treatment based on CT or PET-CT scans, and endoscopy with biopsies.
Duration of response | From date of first CR/PR to the date of first PD according to RECIST criteria, assessed up to 36 months.
  From the date of first CR/PR to the date of first PD.
Treatment-related adverse events | From date of enrollment to the date of last follow-up, assessed up to 36 months.
  Incidence of treatment-related adverse events as assessed by CTCAE v4.0.

OTHER OUTCOMES:
Correlation between immune signature and overall survival | From date of enrollment to the date of last follow-up, assessed up to 36 months.
  The correlation between pretreatment immune signature (PD-L1, CD8, CTLA-4, CD56, and CD68) by mIHC and overall survival.
Correlation between serum cytokines and overall survival and immune-related adverse events | From date of enrollment to the date of last follow-up, assessed up to 36 months.
  The correlation between dynamic change of serum cytokines (IL-2R, IL-6, IL-13, IL-8, CCL3, CD40, and CD274) during treatment and survival outcomes and immune-related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Mian Xi, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Mian Xi, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhu Y, Wen J, Li Q, Chen B, Zhao L, Liu S, Yang Y, Wang S, Lv Y, Li J, Zhang L, Hu Y, Liu M, Xi M. Toripalimab combined with definitive chemoradiotherapy in locally advanced oesophageal squamous cell carcinoma (EC-CRT-001): a single-arm, phase 2 trial. Lancet Oncol. 2023 Apr;24(4):371-382. doi: 10.1016/S1470-2045(23)00060-8. PMID 36990609
- [Result] Ji Y, Du X, Zhu W, Yang Y, Ma J, Zhang L, Li J, Tao H, Xia J, Yang H, Huang J, Bao Y, Du D, Liu D, Wang X, Li C, Yang X, Zeng M, Liu Z, Zheng W, Pu J, Chen J, Hu W, Li P, Wang J, Xu Y, Zheng X, Chen J, Wang W, Tao G, Cai J, Zhao J, Zhu J, Jiang M, Yan Y, Xu G, Bu S, Song B, Xie K, Huang S, Zheng Y, Sheng L, Lai X, Chen Y, Cheng L, Hu X, Ji W, Fang M, Kong Y, Yu X, Li H, Li R, Shi L, Shen W, Zhu C, Lv J, Huang R, He H, Chen M. Efficacy of Concurrent Chemoradiotherapy With S-1 vs Radiotherapy Alone for Older Patients With Esophageal Cancer: A Multicenter Randomized Phase 3 Clinical Trial. JAMA Oncol. 2021 Oct 1;7(10):1459-1466. doi: 10.1001/jamaoncol.2021.2705. PMID 34351356
- [Result] Liu Y, Zheng Z, Li M, Zhang Y, Zhao F, Gong H, Lin H, Huang W, Chen X, Xu Z, Li X, Liu W, Cui Y, Zheng A, Li B. Comparison of concurrent chemoradiotherapy with radiotherapy alone for locally advanced esophageal squamous cell cancer in elderly patients: A randomized, multicenter, phase II clinical trial. Int J Cancer. 2022 Aug 15;151(4):607-615. doi: 10.1002/ijc.34030. Epub 2022 Apr 27. PMID 35419831
- [Result] Wang X, Han W, Zhang W, Wang X, Ge X, Lin Y, Zhou H, Hu M, Wang W, Liu K, Lu J, Qie S, Zhang J, Deng W, Wang L, Han C, Li M, Zhang K, Li L, Wang Q, Shi H, Yu Z, Zhao Y, Sun X, Shi Y, Pang Q, Zhou Z, Liang J, Chen D, Feng Q, Bi N, Zhang T, Deng L, Wang W, Liu W, Wang J, Zhai Y, Wang J, Chen W, Chen J, Xiao Z; Jing-Jin-Ji Esophageal and Esophagogastric Cancer Radiotherapy Oncology Group (3JECROG). Effectiveness of S-1-Based Chemoradiotherapy in Patients 70 Years and Older With Esophageal Squamous Cell Carcinoma: A Randomized Clinical Trial. JAMA Netw Open. 2023 May 1;6(5):e2312625. doi: 10.1001/jamanetworkopen.2023.12625. PMID 37195667